CLINICAL TRIAL: NCT01628679
Title: Physiotherapy Intervention for Provoked Vulvar Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Marcy Dayan, Registered Physiotherapist, Clinical Instructor Department of PhysicalTherapy, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-01805; H11-01805
Record Dates: First submitted 2012-02-12; First posted 2012-06-27 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Vulvodynia; Provoked Vulvar Vestibulodynia
Keywords: provoked; vulvar; vestibulodynia; vestibulitis
MeSH Terms: conditions — Vulvodynia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physical therapy treatment (Experimental)
  Interventions: Behavioral: Physical therapy treatment

INTERVENTIONS:
Behavioral: Physical therapy treatment — Subjects will be given pelvic floor motor control,proprioception and relaxation exercises. This will be with and without the use of external surface Electromyography (EMG) biofeedback. Education will also be given on pain management, female sexual response and vestibulodynia. Subjects will also practice inserting vaginal inserts of graduating diameter into their vaginas, practicing the skills learned in physical therapy sessions.

SUMMARY:
Hypothesis:

1. Specific physiotherapy interventions will decrease pain, improve pelvic floor motor control, increase self efficacy, improve sexual function and decrease pain catastrophizing behaviour in women with provoked vulvar vestibulodynia.

   This study will look at specific physiotherapy treatment interventions to see if they decrease pain, improve pelvic floor motor control, increase self efficacy, improve sexual function and decrease pain catastophizing behaviour. Participants will fill out a questionnaire on their pain symptoms and complete standardized scales prior to starting treatment and after 4 sessions to determine change due to interventions.
2. A combination of physiotherapy, group educational sessions and group cognitive behavioural therapy will have better outcomes than physiotherapy alone.

Results of physiotherapy intervention alone will be compared to results of those treated with physiotherapy, group educational sessions and group cognitive behavioural therapy at a separate treatment centre. Physiotherapy interventions and outcome measures are the same between both groups.

Justification:

Standard treatment is hard to identify as many approaches are taken, none with any evidence to support them. This study aims to look at specific techniques (pelvic floor coordination and relaxation exercises, education on female sexual response and pain pathophysiology education) to see if there is a benefit.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and under
* diagnosis of provoked vulvar vestibulodynia

Exclusion Criteria:

* early menopause
* have had a total or partial hysterectomy
* are on estrogen suppression medication
* have a primary arousal disorder
* declined admission to the Multidisciplinary Vulvodynia Program at Vancovuer General Hospital

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Upon completion of data analysis, establishment of the efficacy of pelvic floor physiotherapy for the treatment of Provoked Vulvar Vestibulodynia will be determined | 2 years
  Time frame: Following completion of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Marcy L Dayan, BSc Rehab, Principal Investigator — Clinical Instructor, Dep't of Physical Therapy, Faculty of Medicine, University of British Columbia
Locations (1):
- Dayan Physiotherapy and Pelvic Floor Clinic, Vancouver, British Columbia, Canada